CLINICAL TRIAL: NCT02443051
Title: Attention Training for Adolescents With Social Anxiety Disorder
Brief Title: Treatment of Social Anxiety in Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Thomas H. Ollendick, Professor - Principal Investigator, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-180THO
Record Dates: First submitted 2015-05-02; First posted 2015-05-13 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Attention Bias Modification (Experimental): Training in bias modification for 80% of experimental trials
  Interventions: Behavioral: Attention Bias Modification
- Control (Active Comparator): Bias modification for 50% of trials
  Interventions: Behavioral: Attention Bias Modification

INTERVENTIONS:
Behavioral: Attention Bias Modification — Computer delivered modification in 80% of trials

SUMMARY:
This research is designed to determine the effectiveness of attention bias modification for socially anxious children and adolescents. Over the course of 3 years, 50 youth will be enrolled in the trial.

DETAILED DESCRIPTION:
The primary objective of this study is to develop an Attention Training (AT) protocol for adolescents with social anxiety disorder (SAD). Attentional biases to threat have been shown to be associated with the development and maintenance of anxiety disorders, in both adults and youth. Given these relations, AT paradigms have been developed to modify these attentional biases. Such paradigms have been shown to be promising in the treatment of adult anxiety. However, to date, only two small studies have examined the use of AT with children, and no ATT protocol has been developed specifically for use with children or adolescents. This is important, given the complications and possible ineffectiveness of applying adult-designed therapies to youth. Given this gap in the literature, the primary aims of the current study are intended to develop a treatment program to address attentional biases and anxiety in adolescents with SAD, to collect preliminary data regarding the program's short-term efficacy and feasibility, and to explore attention biases as a mediator and moderator of initial treatment outcomes. It is hypothesized that the AT protocol developed in the current project, compared to a placebo control comparator condition, will result in reductions in social anxiety among a sample of adolescents with SAD. Further, the AT protocol is expected to reduce attentional biases to threat among those adolescents who possess such biases prior to treatment (not all adolescents are expected to show this bias yet AT has been shown to be potentially effective with these youth; the presence/absence of attention bias will be explored as a moderator of change). The proposed study will be a pivotal step towards assessing the feasibility of an adolescent-focused AT procedure for the treatment of SAD. Results will contribute to an emerging body of research exploring the ameliorating effects of experimental paradigms that target information processing biases in anxious youth. Given emerging evidence regarding the use of AT in adult populations, findings from this study may have implications for improving the current prevention and treatment options available for anxious adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Social Anxiety Disorder;
* English Speaking

Exclusion Criteria:

* Suicide Intent,
* Psychosis,
* Autism Spectrum Disorder

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2013-05; Primary Completion 2016-05 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Clinician Severity Rating | Post-treatment
  Immediately following treatment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas H. Ollendick, Ph.D., Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Child Study Center, Blacksburg, Virginia, United States